CLINICAL TRIAL: NCT03109613
Title: Selecting PEEP in Ventilated Premature Infants by Reducing Ventilation/Perfusion Mismatch: a Pilot Feasibility Study
Brief Title: PEEP and V/Q Mismatch in Premature Infants
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Inadequate enrollment
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-013702
Record Dates: First submitted 2017-04-06; First posted 2017-04-12 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Respiratory Insufficiency Syndrome of Newborn; Infant, Premature, Diseases
Keywords: Positive end-expiratory pressure; PEEP; Bronchopulmonary Dysplasia; Ventilator Induced Lung Injury; V/Q mismatch
MeSH Terms: conditions — Infant, Premature, Diseases; Bronchopulmonary Dysplasia; Ventilator-Induced Lung Injury | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Positive end-expiratory pressure (PEEP) level changes (Experimental): Sequential changes in PEEP level within range of 4-8 cm H2O followed by measurement of V/Q mismatch at each level.
  Interventions: Device: Positive end-expiratory pressure (PEEP)

INTERVENTIONS:
Device: Positive end-expiratory pressure (PEEP) — level changes as per arm description

SUMMARY:
Positive end-expiratory pressure (PEEP) is used in premature infants receiving mechanical ventilation to maintain lungs open and facilitate gas exchange. When ventilation/perfusion mismatch is present, areas of the lung that are open for gas exchange do not match up with areas of the lung that are receiving blood for gas exchange. This study measures the feasibility of enrolling and completing study maneuvers in premature infants for a prospective study measuring the responsiveness of V/Q mismatch to changes in the amount (or level) of PEEP.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm birth before 32 weeks gestational age by best obstetric estimate, determined by the clinical obstetric team during antepartum admission
2. Birth weight less than 1500 grams, as measured by the clinical team at neonatal admission.
3. Presence of endotracheal intubation and invasive mechanical ventilation
4. Less than or equal to 28 days chronologic age
5. Supplemental oxygen requirement, with a fraction of inspired oxygen (FiO2) equal to or greater than 0.25 as documented on the bedside infant flow sheet.

Exclusion Criteria:

1. Congenital anomalies, as determined by the clinical supervising physician
2. Current of prior air leak syndrome, as determined by the clinical supervising physician.
3. Non-English speaking parents
4. Non-viable birth, as determined by the clinical supervising physician

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2016-04-11 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2018-08-08 (Actual)

PRIMARY OUTCOMES:
Feasibility assessed by rate of successfully study enrollment and completion | Full enrollment (12 subjects)
  Rate of successfully study enrollment and completion

SECONDARY OUTCOMES:
Ventilation/perfusion mismatch | 10-20 minutes following each PEEP level change
  Measured by non-invasive computerized technique based of curvilinear characteristics generated by a best-fit curve connection the fractional inspired oxygen and corresponding peripheral oxygen saturation pairs

CONTACTS AND LOCATIONS:
Overall Officials: Haresh Kirpalani, BM, MSc, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Christiana Care Health System, Newark, Delaware
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No